CLINICAL TRIAL: NCT06023329
Title: Superficial Cervical Plexus Block for Improved Outcomes in Pediatric Otolaryngologic Surgery
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: The current PI is leaving the study. Study team is awaiting FDA PI change approval.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ANES-2023-31691
Record Dates: First submitted 2023-08-08; First posted 2023-09-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Otolaryngologic Surgery
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental)
  Interventions: Drug: ropivacaine
- Group 2 (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: ropivacaine — will receive SCPB with ropivacaine via regional anesthesia team
  Arms: Group1
Drug: Saline — will receive SCPB with saline via regional anesthesia team
  Arms: Group 2

SUMMARY:
Literature on the use of superficial cervical plexus blocks for ear surgery is sparse in general, and almost non-existent in the pediatric population. Overall, literature review supports the safety of performance of this block but there is minimal published literature on its utility despite anecdotal evidence of benefit. This study, especially its prospective randomized nature will allow for expansion of the evidence for or against addition of this block to the care of pediatric patients undergoing ear surgery. The purpose of this study is to determine if SCPB plus standard practices provides superior pain control, as measured by reduced opiate consumption, compared to standard practices alone when performed on pediatric patients undergoing surgery on the ear and mastoid process.

ELIGIBILITY:
Inclusion Criteria:

* Age: <18 years and >3 months
* Surgical procedure: Unilateral cochlear implant or tympanomastoidectomy

Exclusion Criteria:

* Preoperative opiate use within the last 30 days
* Bilateral surgery
* No English speaking caregiver
* Parental/patient refusal
* Severe preoperative respiratory compromise
* Allergy to ropivacaine
* Coagulopathy: Defined by INR>1.5 or Platelet count <100k
* Current Infection at site of injection
* VP Shunt on side of surgical procedure
* Pregnant patients: determined by patient history and available laboratory data. Patients will not be required to have pregnancy testing done if not otherwise indicated.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Opioid use | 30 days post surgery
  measured on a MME per kilogram

SECONDARY OUTCOMES:
intraoperative opiate use | 30 days post surgery
  Assessed via chart review of opiate administration on an MME basis
post-operative opiate use | 30 days post surgery
Pain level | 30 days post surgery
  Pain level will be assessed via total pain scores via either FLACC or Wong-Baker Faces, both are pain scales from 0-10, 0 being no pain and 10 being the worst pain imaginable. These scales are interchangeable and will allow both patients who can read and younger patients who cannot read to rate their pain.
Quality of Recovery | 30 days post surgery
  Assessed via modified version of the quality of recovery survey. The quality of recovery scale is a validated document for assessing recovery after surgery. The study will use a modified version of this with language changed for parental assessment of Quality of recovery, but the same questions and scale are used.
Post Anesthesia Care Unit anti-emetic use | 30 days post surgery
  Assessed via chart review of post-operative care unit medication administration

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Fuller, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States